CLINICAL TRIAL: NCT06264518
Title: Exploration of Traumatic Brain Injury Clinical Trials: Unveiling Patient Participation Patterns
Brief Title: An Observational Exploration of Clinical Trials Targeting Traumatic Brain Injury
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 56168915
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical study participation has historically been heavily biased toward specific demographics.

Several people will be invited to enroll in this study so that it may collect a variety of data about traumatic brain injury clinical trial experiences and identify barriers to participation as well as the causes of participants' failure or withdrawal.

People with traumatic brain injury who are invited to take part in medical research will benefit from the analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with traumatic brain injury
* Patient has self-identified as planning to enroll in an observational clinical trial
* Patient is a minimum of 18 years or older

Exclusion Criteria:

* Pregnant or nursing patients
* Inability to perform regular electronic reporting
* Patient does not understand, sign, and return consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Quantity of participants in traumatic brain injury study who sustain participation until study completion
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to enroll in a traumatic brain injury clinical trial | 3 months
Rate of patients who remain in traumatic brain injury clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Giner J, Mesa Galan L, Yus Teruel S, Guallar Espallargas MC, Perez Lopez C, Isla Guerrero A, Roda Frade J. Traumatic brain injury in the new millennium: new population and new management. Neurologia (Engl Ed). 2022 Jun;37(5):383-389. doi: 10.1016/j.nrleng.2019.03.024. Epub 2021 Apr 29. PMID 35672125
- [Background] Hagos A, Tedla F, Tadele A, Zewdie A. Pattern and Outcome of Traumatic Brain Injury, Addis Ababa, Ethiopia: A Cross-sectional Hospital-based Study. Ethiop J Health Sci. 2022 Mar;32(2):343-350. doi: 10.4314/ejhs.v32i2.15. PMID 35693562
- [Background] Shrestha A, Paudel N, Adhikari G, Shrestha S, Lamichhane S, Subedi S, Jaishwal N. Traumatic Brain Injury among Patients Admitted in Neurosurgical Unit in a Tertiary Care Centre: A Descriptive Cross-sectional Study. JNMA J Nepal Med Assoc. 2023 Jun 1;61(262):514-518. doi: 10.31729/jnma.8197. PMID 37464844

DOCUMENTS (1):
  • Informed Consent Form (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT06264518/ICF_000.pdf